CLINICAL TRIAL: NCT05170945
Title: Early Routine Bowel Preparation for Suspected Acute Diverticular Bleeding: A Quality Improvement Initiative Analyzing Hospital Length of Stay
Brief Title: Early Routine Bowel Preparation for Suspected Acute Diverticular Bleeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 003.GID.2020.D
Record Dates: First submitted 2020-09-22; First posted 2021-12-28 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Diverticular Bleeding
MeSH Terms: conditions — Diverticular Diseases | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrospective Cohort (No Intervention): Colonoscopy was performed, either early bowel preparation, late bowel preparation or no bowel preparation patients.
- Prospective Cohort (Experimental): Early bowel preparation for colonoscopy patients
  Interventions: Other: Early bowel preparation for colonoscopy

INTERVENTIONS:
Other: Early bowel preparation for colonoscopy — Early (<24 hours) bowel cleansing prior to colonoscopy.
  Arms: Prospective Cohort

SUMMARY:
This investigation will utilize both a five-year retrospective analysis and a two-year prospective investigation. Variables including age; gender; presence of anticoagulation medication; hospital length of stay; total transfused red blood cell units; presence of heart failure, chronic kidney disease, or lung disease; history of diverticular disease; whether colonoscopy was performed; if therapeutic hemostasis was performed during colonoscopy; and information regarding prior colonoscopies in the past 10 years will be collected for analysis. A small number of early bowel preparation patients are expected in the retrospective study; therefore, a prospective study occurring over the next 12 months will be conducted. Patients agreeing to participate in the study would have a four-liter dose of PEG 3350 ordered, and the medication would be delivered within the first 24 hours of hospitalization. Radiographic studies including computed tomography angiography, tagged RBC scan, and angiography will not be obtained in the first 24 hours of hospital admission and be considered only if the patient has ongoing hematochezia at the completion of their bowel preparation. After completion of the 12-month investigative period (or earlier if sufficient sample size is obtained for clinical significance), data will be analyzed for dissemination consideration.

DETAILED DESCRIPTION:
This investigation will utilize both a five-year retrospective analysis and a two-year prospective investigation. Patient cohorts and data will be obtained through utilization of the EPIC electronic medical record (EMR) and generating an individualized report to capture all possible patients. The report will include all admitted patients with a consult note written by the gastroenterology consult service at Methodist Dallas Medical Center. The consult note will be reviewed, and any patient not meeting the inclusion criteria or those meeting any of the exclusion criteria will be excluded. The patients remaining after this assessment will be included in the retrospective analysis. Variables including age; gender; presence of anticoagulation medication; hospital length of stay; total transfused red blood cell units; presence of heart failure, chronic kidney disease, or lung disease; history of diverticular disease; whether colonoscopy was performed; if therapeutic hemostasis was performed during colonoscopy; and information regarding prior colonoscopies in the past 10 years will be collected for analysis. A small number of early bowel preparation patients are expected in the retrospective study; therefore, a prospective study occurring over the next 12 months will be conducted. The gastroenterology consult service will assess patients with lower GI bleeding with the inclusion and exclusion criteria. Those who qualify will be provided informed consent forms and offered the opportunity to enroll in the study. Patients agreeing to participate in the study would have a four-liter dose of PEG 3350 ordered, and the medication would be delivered within the first 24 hours of hospitalization. Radiographic studies including computed tomography angiography, tagged RBC scan, and angiography will not be obtained in the first 24 hours of hospital admission and be considered only if the patient has ongoing hematochezia at the completion of their bowel preparation. The study is not evaluating effects of colonoscopy, and so any additional intervention performed by the attending gastroenterologist will be subject to their own discretion after the completion of the bowel preparation. After discharge, patient information and data variables will be collected from the EPIC EMR and included in an Excel document. After completion of the 12-month investigative period (or earlier if sufficient sample size is obtained for clinical significance), data will be analyzed for dissemination consideration. Disclaimer: Any cost associated with the procedures stated herein will be billed directly to insurance (as applicable).

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to Methodist Dallas Medical Center
* Age greater than 18 years
* Patient evaluated by gastroenterology consult service during admission
* Hospitalization with diagnosis of "hematochezia", "acute gastrointestinal bleeding", "acute blood loss anemia", or "anemia"
* Endorsed or witnessed episode of painless hematochezia
* Patients exhibiting hemodynamic stability (heart rate <110; systolic blood pressure >90) after initial evaluation and resuscitation by admitting/emergency room physicians

Exclusion Criteria:

* Age less than 18 years
* Persistent hypotension despite initial intravenous fluid resuscitation or fever
* Bowel preparation started 24 hours after initial presentation
* Documented symptoms of dysphagia or odynophagia
* Signs or symptoms suggestive of gastrointestinal obstruction (or ileus) on initial presentation (e.g., abdominal pain, nausea and/or vomiting)
* Inability to complete bowel preparation
* Personal history of inflammatory bowel disease or cirrhosis
* History of immunosuppression (e.g., AIDS, immunosuppressive medication)
* Personal history of colon cancer
* Prior gastric bypass, small bowel, or colonic resection
* Stool culture positive for tested organisms to include Clostridium difficile

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Hospital length of stay | 5 years of data will be collected
  Hospital length of stay in the early bowel preparation, late bowel preparation, and no bowel preparation groups.

SECONDARY OUTCOMES:
Units of RBC transfused | 5 years of data will be collected
  The difference in average units of packed red blood cells transfused during the hospital stay between early, late, and no preparation groups.
Colonoscopy details | 5 years of data will be collected
  Whether a colonoscopy was performed during hospitalization, the diagnosis at time of colonoscopy, and presence of anticoagulation medications.
Therapeutic Hemostasis Invervention | After discharge
  • If a colonoscopy was performed, was therapeutic hemostasis intervention performed.
Radiographic Studies | 5 years of data will be collected
  Number and type of radiographic studies performed to identify source of bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Kedia, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States